CLINICAL TRIAL: NCT04643145
Title: Optimal Drainage After Flexible Ureterorenoscopy; Prospective Assessment of Perioperative Outcomes and Health-Related Quality of Life Through a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AE 201121
Record Dates: First submitted 2020-11-21; First posted 2020-11-24 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Stones, Kidney
Keywords: Kidney stones; Flexible ureteroscopy; Quality of life; drainage
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ureteral catheter (Active Comparator): This group will receive ureteral catheter for 2 days after the procedure
  Interventions: Procedure: Flexible ureteroscopy for renal calculi less than 20 mm
- Indwelling double J stent (Active Comparator): This group will receive indwelling double J stent for 2-4 weeks after the procedure
  Interventions: Procedure: Flexible ureteroscopy for renal calculi less than 20 mm

INTERVENTIONS:
Procedure: Flexible ureteroscopy for renal calculi less than 20 mm — Patients with renal calculi less than 20 mm will be managed by flexible ureteroscopy. at the end of the procedure, they will be randomized to receive either temporary ureteral catheter for 2 days or indweeling double J stent for 2-4 weeks

SUMMARY:
Flexible ureterorenoscopy (FURS) is now recommended for the treatment of kidney stones smaller than 20 mm, as an alternative to extracorporeal shock wave lithotripsy (ESWL) and in combination with percutanous nephrolithotomy (PCNL) for stones larger than 20 mm. At the end of the operation, a ureteral drainage is put in place for the treatment of residual fragments and the inflammation following the ureteroscopy. It helps prevent obstructive symptoms and the development of strictures.

Drainage is done either by a ureteral catheter or by a double J stent. In the literature, while drainage after ureteroscopy is recommended, the criteria for choosing between these two options are not clearly defined.

The objective of this study will be to assess whether the type of postoperative drainage after URS for kidney stones can influence the perioperative outcomes and health-related quality of life.

DETAILED DESCRIPTION:
Flexible ureterorenoscopy (FURS) is now recommended for the treatment of kidney stones smaller than 20 mm, as an alternative to extracorporeal shock wave lithotripsy (ESWL) and in combination with percutanous nephrolithotomy (PCNL) for stones larger than 20 mm. At the end of the operation, a ureteral drainage is put in place for the treatment of residual fragments and the inflammation following the ureteroscopy. It helps prevent obstructive symptoms and the development of strictures.

Drainage is done either by a ureteral catheter or by a double J stent. In the literature, while drainage after ureteroscopy is recommended, the criteria for choosing between these two options are not clearly defined.

The objective of this study will be to assess whether the type of postoperative drainage after URS for kidney stones can influence the perioperative outcomes and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1- Adult patients (aged >18 years) 2- Undergo unilateral uncomplicated retrograde intrarenal surgery (RIRS) using flexible ureterorenoscopy.

Exclusion Criteria:

1. Residual ureteral or renal stones after the procedure as documented by the surgeon
2. Patients who will need auxiliary procedures (ESWL , re-FURS or PCNL)
3. Preoperative febrile UTI
4. pregnancy or breastfeeding
5. Bilateral ureteroscopic surgery
6. Single kidney
7. Chronic kidney disease
8. Cardiovascular or cerebrovascular disease
9. Hepatic dysfunction
10. Other acute medical conditions as acute gastroenteritis, osetoarthritis that might influence the patient QoL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 12 weeks after the procedure
  presence of residual fragments on non contrast computed tomography

SECONDARY OUTCOMES:
perioperative complications | First 3 days postoperative
  perioperative complications after the procedure
Postoperative pain by visual analogue scale | first 24 hours postoperatively
  Visual analogue scale will be assessed postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt